CLINICAL TRIAL: NCT03729947
Title: CLOSED SUCTION DRAIN VS. NO DRAIN IN ADOLESCENTS UNDERGOING PEDICLE SCREW INSTRUMENTATION FOR IDIOPATHIC SCOLIOSIS (DAISY 2018). A Randomized Clinical Trial
Acronym: DAISY 2018
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Karolinska Institutet (Other); Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Ilkka Helenius, Professor of Pediatric Orthopedics, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 95/2018
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drain placed (Active Comparator): Subfascial drain at end of procedure
  Interventions: Device: Subfascial closed suction drain
- No drain placed (Placebo Comparator): No drain left at the end of study
  Interventions: Device: Subfascial closed suction drain

INTERVENTIONS:
Device: Subfascial closed suction drain — Ch 14 closed suction drain
  Other Names: No other

SUMMARY:
Abstract Background - Closed suction drain is typically used worldwide after instrumented posterior spinal fusion for adolescent idiopathic scoliosis (AIS). Postoperative drain leakage has been associated with up to 50% of total blood loss in these patients. Previous studies on adult patients with degenerative lumbar spine disorders have shown that leaving out subfascial drain does not increase the risk of deep wound infection or epidural hematoma. However, there has been no studies evaluating the need for subfascial drain in adolescents undergoing instrumented spinal fusion for idiopathic scoliosis.

Study Design - A randomized, multicenter clinical trial on children and adolescents undergoing posterior spinal fusion for idiopathic scoliosis using pedicle screw technique. Ninety consecutive adolescents will be randomized into drain vs. no drain group at the time of wound closure using the sealed envelope technique (1:1).

Aims and hypothesis - To compare drain vs. no drain use groups for the change in postoperative hemoglobin or hematocrit in children undergoing posterior spinal fusion for AIS. We hypothesize that postoperative hemoglobin change will be larger in the group receiving subfascial drain and there will no change in the risk of postoperative complications (deep surgical site infection, need for hematoma evacuation or other re-operation) between the study groups.

Inclusion criteria - Adolescents (aged 10 to 21 years of age) undergoing surgery for idiopathic scoliosis using pedicle screw technique.

Exclusion criteria - Coagulation disorder, smoking, unwilling to consent, vertebral column resection, need for anteroposterior surgery.

Main outcome parametres - Postoperative change in hemoglobin or hematocrit; Secondary parametres: need for blood transfusion, need for re-operation, need for change in the dressings.

Ethical aspects - Ethical committee approval will be obtained both in Finland and in Sweden. An informed consent will be obtained from all children and their parents. In case of major intraoperative blood loss (>50% of blood volume) a subfascial drain can be inserted based on the decision of the treating physician.

Time schedule and budget - This study will be started after ethical committee approval (estimated 10/2018). There will be no extra costs as all information gathered will be part of normal surgical treatment of AIS. A part-time research nurse has been hired to take care of data collection into the database.

DETAILED DESCRIPTION:
Background The use of a subfascial closed suction drain has been a long tradition in adolescents undergoing posterior spinal fusion for idiopathic scoliosis.1-5 Drain has been used to limit postoperative hematoma and epidural hematoma formation, to decrease risk of postoperative deep wound infection, and to shorten hospital stay. Postoperative 24 hour drain output has been larger than introperative blood loss in these patients.6 Previous studies in adults undergoing total joint replacement have shown increased risk of hematocrit decrease and blood transfusion, but better joint mobilization in patients treated with closed suction drain as compared with those not receiving drain. In patients with lumbar degenerative disorders drain use has been associated with higher risk of blood transfusion and longer hospital stay.7-8 Leaving out subfascial drain has not been associated with increased risk of deep surgical site infection or neurologic deficit, but the number of patients with postoperative saturated dressings has been larger.1-5 There are no Level 1 studies evaluating the need to use a subfascial closed suction drain or not in adolescents undergoing posterior spinal fusion for idiopathic scoliosis.

Aims and hypothesis To compare postoperative Hemoglobin and hematocrit decrease, length of hospital stay, and hematoma formation in patients receiving and not receiving subfascial drain during posterior spinal fusion for idiopathic scoliosis. We hypothesize that children not receiving a subfascial drain demonstrate smaller hemoglobin and hematocrit decrease without increased risk of wound or neurologic complications.

Methods Study design - A randomised, multicentre clinical trial according to CONSORT criteria.9 Patients - 90 adolescents undergoing posterior spinal fusion with pedicle screw instrumentation for idiopathic scoliosis will be randomized at the time of wound closure receiving a single subfascial drain (Hemovac 14 ch) or no drain.

Inclusion criteria - Patients will be included if they fulfilled the following criteria: between ten and 21 years of age; no contraindication to the use of subfascial drain; suitable for posterior scoliosis surgery using all pedicle screw technique for AIS (Lenke classification10 Types 1 to 6); normal blood coagulation; a normal whole spine MRI except for the spinal deformity (juvenile or AIS). Exclusion criteria - Need for anteroposterior surgery; the need for vertebral resection; smoking; diabetes mellitus or abnormalities in blood coagulation. Use of non-steroidal anti-inflammatory should be avoided within one week of surgery.

Intervention - The intervention group will receive a single subfascial drain (Hemovac Ch14; Zimmer, Warsaw, Indiana). The control group will not receive a drain.

Randomization - Randomization to intervention and control groups (1:1) will be carried out using the sealed envelope technique at the time of wound closure.

Outcomes - The main outcome measures include postoperative decrease in hemoglobin, hematocrit and the need for blood products (packed red cells, frozen plasma or platelets). Secondary outcome measures include blood loss (mls), drain output over 24 hours (mls), total blood loss (intra-operative blood loss + drain output); 48 hour opioid consumption (mg/kg); body temperature during postoperative hospital stay; the number of patients with fully saturated wound dressings requiring exchange will be recorded.

Surgery - Surgical planning of implant placement and the need for the Ponte procedure will be carried out preoperatively. Each patient will be placed in the prone position and the posterior elements will be exposed using electrocautery. The deformity will be corrected using bilateral segmental pedicle screw instrumentation and en bloc vertebral column derotation. Spinal fusion is carried out using autograft acquired from facetectomies and osteotomies with bone graft extenders (Grafton, Medtronics Spinal and Biologics). Spinal cord monitoring (MEP, SSEP, lumbar nerve root EMG with or without pedicle screw stimulation) will be undertaken in all patients. A single subfascial drain (Hemovac Ch14; Zimmer, Warsaw, Indiana) will be placed according to randomization during closure and will be removed at 24 hours post-operatively. A sterile wound dressing will be applied at the end of surgery. Wound dressings will not be changed before discharge, until they are fully saturated.

Anaesthesia - All patients will have total intravenous anesthesia including dexmedetomidine, propofol and remifentanil with the aim of achieving a mean arterial pressure between 65 mmHg and 75 mmHg during surgery and for the first 24 hours post-operatively. Cefuroxime and Vancomycin will be used as antibiotic prophylaxis.

All patients will receive an intravenous bolus of tranexamic acid (30 mg/kg, maximum dose 1500 mg) within 30 minutes before incision and then an infusion (10 mg/kg/h, maximum dose 500 mg/h) during surgery. Intra-operative blood loss will be measured and recorded as the amount of blood collected in the cell saver, surgical wound dressings will be weighed during surgery, excluding any irrigation with saline. The cell saver will be used in all patients and the amount of autologous blood returned is recorded. Allogenic red blood cells will be transfused if the Hb concentration goes below 80 g/L during surgery or during the hospital stay. Fresh frozen plasma will be given if the blood loss exceeds 50% of the patients total blood volume. Platelets will be infused if the blood loss is more than 100% of the blood volume. The estimated blood volume will be calculated using a formula of 70 ml/kg x weight (kg).12 Statistical power - The sample-size requirement of 30 patients per group was calculated using a study power of 80%, a type I error (alpha) of 0.05, and an estimated effect size of 0.7. Effect size evaluation was based on the assumption that mean (SD) postoperative hemoglobin loss (the primary endpoint) would be 30 g/l (SD 14) for the control group and 40 (SD 14) for the intervention group.6 We further expand the sample size calculation by 16% to adjust the results for possible non-parametric methods. To accommodate for possible drop outs during the follow-up 90 patients will be enrolled.

Ethical aspects Ethical committee approval will be obtained at our university hospital. If the subfascial drain could not be used e.g. due to cerebrospinal fluid leakage or based on the surgeon's judgment, leaving it will be allowed, however, the patient will remain in the intervention group for statistical comparison according to the intention-to-treat principle.

Time schedule This study will be started after ethical committee approval estimated in the beginning of 2019 and patient recruitment is estimated to be done by the end of 2023.

Budget Surgical treatment of adolescents with idiopathic scoliosis is according to the standard practice. There will be no extra costs due to this study. A part-time research nurse and PhD students will be hired using Valtion tutkimusrahoitus and external funding.

References

1. Brown MD, Brookfield KF. A randomized study of closed wound suction drainage for extensive lumbar spine surgery Spine (Phila Pa 1976). 2004 May 15;29(10):1066-8.
2. Kanayama M, Oha F, Togawa D, Shigenobu K, Hashimoto T. Is closed-suction drainage necessary for single-level lumbar decompression?: review of 560 cases. Clin Orthop Relat Res. 2010 Oct;468(10):2690-4.
3. Zijlmans JL, Buis DR, Verbaan D, Vandertop WP. Wound drains in non-complex lumbar surgery: a systematic review. Bone Joint J. 2016 Jul;98-B(7):984-9.
4. Liu Y, Li Y, Miao J. Wound drains in posterior spinal surgery: a meta-analysis. J Orthop Surg Res. 2016 Jan 22;11:16.
5. Liu JM, Chen WZ, Fu BQ, Chen JW, Liu ZL, Huang SH. The Use of Closed Suction Drainage in Lumbar Spinal Surgery: Is It Really Necessary? World Neurosurg. 2016 Jun;90:109-115.
6. Helenius I, Keskinen H, Syvänen J, Lukkarinen H, Mattila M, Välipakka J, Pajulo O. Gelatine matrix with human thrombin decreases blood loss in adolescents undergoing posterior spinal fusion for idiopathic scoliosis. A MULTICENTRE, RANDOMISED CLINICAL TRIAL. Bone Joint J 2016;98-B:395-401.
7. Parker MJ, Roberts CP, Hay D. Closed suction drainage for hip and knee arthroplasty. A meta-analysis. J Bone Joint Surg Am. 2004 Jun;86-A(6):1146-52
8. Zhang Q, Liu L, Sun W, Gao F, Zhang Q, Cheng L, Li Z. Are closed suction drains necessary for primary total knee arthroplasty?: A systematic review and meta-analysis. Medicine (Baltimore). 2018 Jul;97(30):e11290
9. Schulz KF, Altman DG, Moher D, CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ 2010;340:332.
10. Mattila M, Jalanko T, Helenius I. En bloc vertebral column derotation provides spinal derotation but no additional effect on thoracic rib hump correction as compared with no derotation in adolescents undergoing surgery for idiopathic scoliosis with total pedicle screw instrumentation. Spine (Phila Pa 1976) 2013;38:1576-1583.
11. Lenke LG, Betz RR, Harms J, et al. Adolescent idiopathic scoliosis: a new classifi- cation to determine extent of spinal arthrodesis. J Bone Joint Surg [Am] 2001;83- A:1169-1181.

Cote CJ. Pediatric Anesthesia. In: Miller RD, Eriksson LI, Fleisher LA, Wiener-Kronish JP, Young WL, eds. Miller's Anesthesia. Philadelphia: Churchill Livingstone; 2010:2559-2597.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they fulfilled the following criteria: between ten and 21 years of age; no contraindication to the use of subfascial drain; suitable for posterior scoliosis surgery using all pedicle screw technique for AIS (Lenke classification10 Types 1 to 6); normal blood coagulation; a normal whole spine MRI except for the spinal deformity (juvenile or AIS).

Exclusion Criteria:

* Need for anteroposterior surgery; the need for vertebral resection; smoking; diabetes mellitus or abnormalities in blood coagulation. Use of non-steroidal anti-inflammatory should be avoided within one week of surgery.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Postoperative change in Hemoglobin | Postoperative days 1-3
  Hemoglobin
Postoperative pain | Postoperative days 1-3
  Visual analogue scale

SECONDARY OUTCOMES:
Postoperative use of opioids using patient controlled analgesia | Postoperative days 1-2
  Opioid consumption

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka J Helenius, MD, Prof, Principal Investigator — Turku University Hospital
Locations (3):
- Finland (2):
  - Turku University Hospital, Turku
  - Turku Children's Hospital, Turku
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No